CLINICAL TRIAL: NCT04604418
Title: Outcomes and Health Care Resource Utilization in Pediatric Congenital Heart Disease Patients Undergoing Non-Cardiac Procedures
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: The Hospital for Sick Children (Other); Vanderbilt University Medical Center (Other); University of Minnesota (Other); Children's Hospital of Philadelphia (Other); Children's Healthcare of Atlanta (Other); Baylor College of Medicine (Other); Children's National Research Institute (Other); Children's Hospital of The King's Daughters (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Viviane Nasr, Associate Professor, Boston Children's Hospital
Other Study IDs: IRB-P00035008
Record Dates: First submitted 2020-10-16; First posted 2020-10-27 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Congenital Heart Disease in Children
Keywords: Perioperative risk prediction; Adverse Postoperative Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention. It is observational — No intervention. It is observational

SUMMARY:
The incidence of moderate to severe congenital heart disease (CHD) in the United States is estimated to be 6 per 1000 live-born full term infants. Recent advances in pediatric cardiology, surgery and critical care have significantly improved the survival rates of patients with CHD leading to an increase in prevalence in both children and adults. Children with CHD significant enough to require cardiac surgery frequently also undergo non-cardiac surgical procedures. Analysis of the Pediatric Health Information System database between 2004 and 2012 demonstrated that 41% of children who had undergone surgery to correct CHD in the first year of life also underwent at least one non-cardiac surgery by age 5. With this increased demand for non-cardiac procedures, anesthesiologists, pediatricians and other healthcare providers will encounter patients with repaired or unrepaired CHD and other cardiac diseases in their practice.

However, the information provided by national databases lack granularity and the information from single institutional data is limited.

This project aims to address this knowledge gap in quantifying the risk for cardiac patients coming for noncardiac procedures and identify the health care resource utilization and system to best care for this patient population. To conduct this study, we will create a multi-institutional collaboration between large and small centers to create a unique dataset spanning all the different variables that need to be considered in risk prediction for these patients including patient variables, hospital setting, and providers. The aggregate multiinstitutional data set may be used for benchmarking for national quality improvement efforts.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages birth to 21 years.
2. Patients diagnosed with congenital heart disease
3. Patients undergoing a noncardiac procedure (surgical or nonsurgical)

Exclusion Criteria:

1. Patients with congenial heart disease undergoing a cardiac surgical procedure including pacemakers.
2. Patients with congenital heart disease undergoing a catheterization(diagnostic or interventional) or an electrophysiology study

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with congenital heart disease and presenting to the participating institution for a noncardiac procedure are included in the study.
  All patients will be included.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | during the procedure and up to 30-days following the procedure
  Death
Intensive Care Unit admission | following the procedure and up to 72 hours
  The postoperative location of the patient is in the intensive care unit unexpectedly
Postoperative mechanical support | following the procedure and up to 72 hours
  Patient required a ventilator or noninvasive positive pressure ventilation
Intraoperative cardiac event | During the perioperative period

SECONDARY OUTCOMES:
Readmission Cardiac arrest: during the procedure and up to 72 hours Neurologic injury (stroke, seizure) following the procedure and up to 72 hours Renal injury following the procedure and up to 72 hours | following the procedure and up to 72 hours
  Patient was discharged after the procedure and needed to be readmitted to the hospital is defined as readmission
Cardiac arrest | during the procedure and up to 72 hours
  Patient required cardiopulmonary ressuscitation
Neurologic injury | Following the procedure and up to 72 hours
  Defined as stroke or seizure by the provider
Renal Injury | Following the procedure and up to 72 hours
  Defined based on creatinine and glomerular filtration

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Nasr, MD, Principal Investigator — Boston Children's Hospital
Locations (10):
- United States (9):
  - University of California, Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston Hospita, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of the King's Daughter, Norfolk, Virginia
- Hospital for Sick Kids, Toronto, Ontario, Canada